CLINICAL TRIAL: NCT02498704
Title: The Effectiveness of Dry Needling and Stretching vs. Stretching Alone on Hamstring Flexibility in Patients With Knee Pain: A Randomized Controlled Trial
Brief Title: Dry Needling and Stretching vs. Stretching Alone on Hamstring Flexibility in Patients With Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, John Mason, Sports Physical Therapy Fellow, Keller Army Community Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 403645-1
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Mobility Limitation
MeSH Terms: conditions — Mobility Limitation | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Needling intervention, Control (Sham Comparator): Sham dry needling, group does not receive true dry needling intervention.
  Interventions: Other: Sham Needling
- Dry Needling Intervention, experimental (Experimental): Group receives true dry needling intervention.
  Interventions: Procedure: Dry Needling

INTERVENTIONS:
Procedure: Dry Needling — Trigger point dry needling to hamstring muscle group.
  Arms: Dry Needling Intervention, experimental
Other: Sham Needling — Superficial palpation of trigger point, skin is not punctured.
  Arms: Sham Needling intervention, Control

SUMMARY:
The purposes of this double-blinded, randomized controlled trial are (1) to determine if the addition of trigger point dry needling (TDN) to a standard stretching program results in greater improvements in hamstring flexibility versus stretching alone in a population with atraumatic knee pain; (2) measure length of time that flexibility gains are maintained, (3) assess resulting movement mechanics and (4) assess patient reported changes in pain. Findings will potentially lead to insights as to the benefit of applying this intervention to additional body regions.

DETAILED DESCRIPTION:
In this study, up to 40 subjects with a history of atraumatic knee pain will be randomized into 2 groups of up to 20 subjects per group (1 experimental group and 1 control group). Subjects in the experimental group will receive TDN intervention with hamstring stretching while subjects in the control group will receive an alternative needling intervention with hamstring stretching. After meeting all inclusion criteria, all subjects will undergo the following tests: supine active knee extension, the active straight leg raise test, deep squat, and a single leg step down from a 6 inch step. Subjects who measure less than 20° from full extension on the active knee extension test will be excluded. Hamstring tightness has been operationally defined as having greater than 20° loss of knee extension as measured with the femur held at 90° of hip flexion.[1] Manual palpation of the bilateral biceps femoris, semitendinosus, and semimembranosus will be performed to detect the presence of myofascial trigger points (TPs) in groups 1 and 2. Dry needling will be performed to all detected TPs by a provider trained and experienced in TDN. Post TDN, all tests will be immediately repeated and at each follow up the subject will complete the Global Rating of Change survey (GROC) and Lower Extremity Functional Scale (LEFS).

Post intervention, subjects in experimental group 1 will be given a standing hamstring stretch to perform 1 repetition held for 30 seconds, repeated 3 times daily. These parameters have been shown to be effective at improving flexibility.[2] Subjects will be instructed by demonstration and will be provided with a handout of stretching instructions. Subjects will be given an exercise log to record home exercise compliance.

Subjects in group 2 will be given an alternative needling intervention followed by a standing hamstring stretch to perform 3 times per day, 1 repetition held for 30 seconds. Alternative needling intervention will be performed to give the appearance of regular TDN intervention; however, no needle penetration will be performed. Following alternative needling intervention, subjects will be instructed by demonstration and will be provided with a handout of hamstring stretching instructions. Home exercise compliance will be recorded at each follow up.

Follow up measurements will be recorded between 1-2 days, 3-4 days, and 7-8 days post intervention. All tests will be repeated. One additional session of TDN and alternative needling intervention will be performed at day 3-4.

ELIGIBILITY:
Inclusion Criteria:

* Department of Defense healthcare beneficiaries
* 18-40 years old
* atraumatic knee pain greater than 2 weeks in duration
* Lack of 20 degrees or more of active supine knee extension

Exclusion Criteria:

* History of herniated lumbar disc/radiculopathy
* Prior surgery in the hip, knee or back
* Self-Reported Pregnancy
* History of blood borne pathogens/infectious disease/active infection/metal allergy
* Knee pain of traumatic origin, instability, joint line tenderness, or positive meniscal tests
* Participants who are not fluent in English
* Previous history of TDN
* Bleeding disorders or currently taking anti-coagulant medications

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Knee extension range of motion | 7-8 days
  Assessed with active supine knee extension and supine straight leg raise using digital inclinometer

SECONDARY OUTCOMES:
knee pain with squat recorded on visual analog scale | 7-8 days
knee pain with step down test recorded on visual analog scale | 7-8 days
lower extremity functional scale (LEFS) | 7-8 days
  Self Report Functional Outcome measure
Global Rating of Change | 7-8 days
  Self Report Functional Outcome measure
knee range of motion during squat | 7-8 days
  knee flexion measured with standard goniometer during squat

CONTACTS AND LOCATIONS:
Overall Officials: John Mason, DPT, Principal Investigator — Keller Army Community Hospital
Locations (1):
- Keller Army Community Hospital, West Point, New York, United States